CLINICAL TRIAL: NCT01450787
Title: Prevalence of Dry Eyes in Diabetics Compared to Non Diabetics
Status: Terminated | Type: Observational
Why Stopped: Principle investigator changed practice location and discontinued study
Sponsor: COA Research Foundation, INC (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: 000322
Record Dates: First submitted 2011-10-10; First posted 2011-10-12 (Estimated); Results first posted 2013-09-30 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-08

CONDITIONS: Dry Eyes
Keywords: dry eyes; diabetes
MeSH Terms: conditions — Dry Eye Syndromes; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- diabetics: diabetics
- non diabetics: non diabetics

SUMMARY:
The purpose is to compare the prevalence of dry eyes in diabetics and non diabetics. This might help identify a group of patients at greater risk for dry eye complications. Diabetics have been shown to have poor ocular surface healing and might benefit from dry eye therapy earlier if they are shown to be at greater risk for dry eyes.

DETAILED DESCRIPTION:
Dry eye disease is one of the most common eye problems seen in ophthalmology. Diabetics are at high risk for multiple eye problems, including retinopathy and glaucoma. They also have been shown to have poor ocular surface healing. I would like to evaluate the prevalence of dry eye disease in diabetics to see if they are also at greater risk for the known complications of dry eye disease. If so, they might benefit from early intervention.

ELIGIBILITY:
Inclusion Criteria:

* 50 patients with diabetes, 25 without diabetes over the age of 40

Exclusion Criteria:

* current use of glaucoma drops or currently within the postoperative period from eye surgery

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Existing clinic population from our practice
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth A Beckman, MD, Principal Investigator — COA Research Foundation
Locations (1):
- Columbus Ophthalmalogy Associates, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled randomly. Consecutive patients in a private ophthalmology clinic that met inclusion criteria were asked to participate at the time of an already scheduled exam. The non-diabetic group recruitment stopped once the target number of subjects enrolled. The diabetic group recruitment continued until the study was terminated.
Pre-assignment Details: Being that there was no intervention and the study only involved taking measurements at the time of the exam, there was no transition required. Any eligible patient that was willing to participate was included. Consecutive diabetic patients and consecutive non-diabetic patients that met criteria were offered the opportunity to enroll.
Groups:
- Diabetics: diabetics over age 40
- Non Diabetics: non diabetics over age 40
Period: Overall Study
Arm/Group | Diabetics | Non Diabetics
Started | 38 | 25
Completed | 38 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diabetics | Non Diabetics | Total
Number analyzed (Participants) | 38 | 25 | 63
Age, Customized [Number; unit: participants] | 38 | 25 | 63
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 43
  Male | 16 | 4 | 20
Region of Enrollment [Number; unit: participants]
  United States | 38 | 25 | 63

OUTCOME MEASURES:

1. Primary Outcome: Conjunctival Staining Score
Description: Conjunctival staining with lissamine green dye is measured at the time of the evaluation on a scale from 0 to 5 using the oxford scoring system, with 5 being the most severe staining.
Time Frame: at the time of the evaluation
Population: There were 38 consecutive diabetics over 40 years of age and 25 consecutive non-diabetics over 40 years of age that qualified and agreed to enroll. A target of 25 non-diabetics was met. The target of 50 was not met as the study was stopped when the PI changed practices. By that time, 38 diabetics enrolled.
Measure: Mean (Standard Error); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Diabetics | Non Diabetics
Number analyzed (Participants) | 38 | 25
Number analyzed (eyes) | 76 | 50
units on a scale | 2.72 (0.16) | 2.19 (0.19)

2. Secondary Outcome: Tear Film Osmolarity
Description: The tear film osmolarity is measured at the time of the exam.
Time Frame: at the time of the exam
Population: Tear film osmolarity was measured in all patients, but two patients in the diabetic group had an insufficient tear film to obtain a reading. Therefore, only 36 diabetics were included.
Measure: Mean (Standard Error); unit: mOsml/L
Units Other Than Participants: eyes
Arm/Group | Diabetics | Non Diabetics
Number analyzed (Participants) | 36 | 25
Number analyzed (eyes) | 72 | 50
mOsml/L | 303.41 (2.03) | 312.06 (3.05)

3. Other Pre Specified Outcome: OSDI Score
Description: The ocular surface disease index survey in completed at the time of the exam. This scale ranges from 0 to 100 higher scores representing greater disability.
Time Frame: at the time of the exam
Population: All patients completed the OSDI survey
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Diabetics | Non Diabetics
Number analyzed (Participants) | 38 | 25
units on a scale | 19.58 (2.62) | 27.50 (4.60)

4. Other Pre Specified Outcome: Schirmer Score
Description: The schirmer tear production test with anesthesia is completed at the time of the exam in mm of tear film absorption on the test strip after five minutes. Higher scores represent greater tear production.
Time Frame: at the time of the exam
Population: Each patient underwent schirmer testing
Measure: Mean (Standard Error); unit: mm
Units Other Than Participants: eyes
Arm/Group | Diabetics | Non Diabetics
Number analyzed (Participants) | 38 | 25
Number analyzed (eyes) | 76 | 50
mm | 18.36 (1.06) | 15.88 (1.34)

5. Other Pre Specified Outcome: Tear Break-up Time
Description: The tear break-up time with fluorescein solution is measured at the time of the exam in seconds.
Time Frame: at the time of the exam
Population: Each patient underwent tear break-up time testing
Measure: Mean (Standard Error); unit: seconds
Units Other Than Participants: eyes
Arm/Group | Diabetics | Non Diabetics
Number analyzed (Participants) | 38 | 25
Number analyzed (eyes) | 76 | 50
seconds | 3.38 (0.17) | 3.66 (0.26)

6. Other Pre Specified Outcome: Corneal Staining
Description: Corneal staining with fluorescein solution is graded at the time of the exam on a scale of 0 to 5 using the oxford scoring system with 5 being the most severe staining.
Time Frame: at the time of the exam
Population: All patients underwent corneal staining evaluations using fluorescein.
Measure: Mean (Standard Error); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Diabetics | Non Diabetics
Number analyzed (Participants) | 38 | 25
Number analyzed (eyes) | 76 | 50
units on a scale | 0.31 (0.08) | 0.30 (0.13)

ADVERSE EVENTS:
Arm/Group | Diabetics | Non Diabetics
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/25
Other Adverse Events (participants affected / at risk) | 0/38 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No